CLINICAL TRIAL: NCT06184867
Title: Choices About Genetic Testing And Learning Your Risk With Smart Technology
Acronym: CATALYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Director at Rutgers Cancer Institute, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 132307; Pro2023000964 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2023-11-07; First posted 2023-12-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Breast Cancer; Pancreas Cancer; Colorectal Cancer; Endometrial Cancer; Prostate Cancer
Keywords: hereditary cancer; genetic testing; genetic education; relational agent; chatbot
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Prostatic Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm parallel-group randomized controlled trial designed to evaluate the feasibility and acceptability of the relational agent/chatbot (RA) intervention versus enhanced usual care (EUC) among cancer survivors. Randomization will occur at the patient level, with a 1:1 ratio. Phase 1 will enroll 8 participants for user testing, Phase 2 will enroll 6 participants for usability testing, and Phase 3 will enroll 36 participants for pilot testing.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Treating clinicians will be blind to their patient's group assignment. While participants cannot be blinded to the group, they will be blinded to the study's specific hypotheses. Statisticians and outcome assessors will be blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relational Agent (RA) (Experimental): Participants in the RA arm will receive a clinical letter signed by the Medical Director of the institution's clinical genetics program with a link to the HIPAA-compliant RA. The RA will provide educational content equivalent to traditional genetic counseling (GC) in a streamlined format, including videos, decision support, patient testimonials, and real-time Q&A. Participants will be informed that they can consult with a genetic risk specialist at no cost. Those opting for genetic testing (GT) will have a kit mailed to them, with results shared with the participant and their oncologist, tailored to the findings. Participants undecided or unwilling to proceed with GT will be encouraged by the RA to consult their oncology provider and/or schedule a GC appointment.
  Interventions: Behavioral: Relational Agent (RA)
- Enhanced Usual Care (EUC) (Active Comparator): Participants in the EUC arm will receive a clinical letter signed by the Medical Director of the institution's clinical genetics program. The letter will inform participants of their and their family's potential risk for carrying a pathogenic variant (PV) associated with hereditary cancer. It will emphasize their eligibility for genetic testing (GT), recommend considering a genetic counseling (GC) appointment for further information, and provide a link to the Rutgers Cancer Institute high-risk clinic website. The study team will assist in facilitating GT upon request. Results will be shared with the participant and their oncologist and tailored according to the findings.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Relational Agent (RA) — Consists of a clinical letter and engagement with genetic education and uptake of genetic testing for hereditary cancer risk among cancer survivors.
  Other Names: Alex; Chatbot; Digital health tool; Decision support tool
  Arms: Relational Agent (RA)
Behavioral: Enhanced Usual Care (EUC) — Consists of a clinical letter and recommendation for genetic testing for hereditary cancer risk among cancer survivors.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study seeks to enhance genetic education and increase the uptake of genetic testing for hereditary cancer risk among cancer survivors. The study will focus on the feasibility and acceptability of a digital intervention designed to improve cancer genomic care.

The study objectives are to:

1. Finalize the development and optimize the usability of the CATALYST digital intervention (also known as the relational assistant [RA]).
2. Evaluate the feasibility and acceptability of a streamlined cancer genomic care delivery model for cancer survivors. Participants will be randomized to one of two study arms: the RA intervention arm or the enhanced usual care (EUC) arm.
3. Assess the uptake of genetic counseling (GC) and genetic testing (GT) and conduct a process evaluation to identify barriers and facilitators to GC, GT, and engagement with the CATALYST intervention and the RA.

DETAILED DESCRIPTION:
Research Design and Methods:

This study encompasses refinement of the digital intervention prototype through usability and user interface testing, and subsequent pilot/feasibility testing of a multi-level intervention, CATALYST, that includes a novel digital cancer genetic risk assistant that incorporates education, decision support, interactive smart technology and provides personalized information regarding hereditary cancer risk and genetic testing. The study will be comprised of three intervention testing stages: Phase 1 - User Testing; Phase 2 - Usability Testing, and Phase 3 - Pilot Testing.

User testing and usability testing will be done to refine the intervention prototype by incorporating cancer patients' feedback during each phase. The feasibility and acceptability of the CATALYST intervention will be evaluated in a 2-armed randomized controlled pilot study (Phase 3) of 36 individuals (18 EUC, 18 RA arm) identified as high-risk for a hereditary cancer gene mutation according to NCCN Criteria. The primary outcome of interest is GT uptake.

Data will be collected via guided interviews (televideo or face-to-face in the clinic or other mutually convenient location (community center) for Phase 1 and Phase 2. Phase 3 surveys will be self-administered via the internet or interviewer administered via telephone. Interviews and surveys will be comprised of open-ended and close-ended questions.

ELIGIBILITY:
Inclusion Criteria:

User/Usability Testing

1. Age 18 or older
2. Diagnosed with ovarian, fallopian tube, peritoneal, breast, pancreatic, colorectal, endometrial or prostate cancer
3. Speak/read and understand English
4. Capable of providing informed consent
5. Have Internet access (via smartphone, tablet, or computer)

Randomized Feasibility Trial

1. Age 18 or older
2. Diagnosed with ovarian, fallopian tube, peritoneal, breast, pancreatic, colorectal, endometrial or prostate cancer
3. Meet National Comprehensive Cancer Network (NCCN) criteria for germline GT
4. Speak/read and understand English
5. Capable of providing informed consent
6. Have Internet access (via smartphone, tablet or computer)

Exclusion Criteria:

Participants will be 18 years of age or older because germline genetic testing is generally not recommended in children when the test results would not impact clinical management. Participants from the user and usability testing phases are not eligible for the feasibility trial. Feasibility trial participants cannot have previously undergone germline GT for hereditary cancer risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Genetic Testing (GT) Uptake | 1-month, 6-month follow-up
  GT uptake will be defined as the proportion of participants who undergo genetic testing within 6 months of the baseline survey (for both the EUC and RA arms). This will be verified through medical record documentation. Self-reported GT will be tracked if verification is not feasible.

SECONDARY OUTCOMES:
Acceptability of the Relational Agent (RA) | 1-month follow-up
  Acceptability will be assessed using the Chatbot Usability Questionnaire (CUQ), which evaluates key aspects of the chatbot, including its personality, onboarding process, user experience, and error handling.
  The CUQ consists of 16 items, each rated on a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree), with scores ranging from 16 to 80. These scores will be normalized to a scale of 100. A CUQ score of 68 or higher will indicate acceptable usability.
Genetic Testing (GT) Intentions | Baseline, 1-month, 6-month follow-up
  GT intentions will be assessed using a single-item question based on the Ottawa Decision Support Framework, with six options that assess participants' readiness to engage in decision-making, ranging from not considering the choices to having already made a decision and being unlikely to change. This operationalization captures the concept of reactance to health messaging, an EPPM construct.
Informed Decision-Making Indicators | Baseline, 1-month, 6-month follow-up
  Hereditary Cancer Knowledge will assess understanding of hereditary cancer, inheritance patterns, risk factors, and genetic testing implications using a 10-item Knowledge Index based on ASCO guidelines. Response options include "Agree," "Disagree," or "I don't know."
  Decision Conflict will be measured with a 12-item scale on uncertainty, being informed, personal values, and support in decision-making, plus 4 items on decision quality. Items are rated on a 5-point Likert scale (Cronbach's alpha = 0.78).
  Decision Regret will be assessed using a 5-item scale on distress/remorse post-decision (Cronbach's alpha = 0.81-0.92).
  Decision Satisfaction will use a 6-item scale (Cronbach's alpha = 0.86).
  Psychological distress will be assessed using the PROMIS anxiety and depression subscales.
  Health Beliefs will assess Perceived Susceptibility, Self-Efficacy for genetic testing, and Response Efficacy using 4 items per subscale (Cronbach's alpha = 0.85-0.93).
Genetic Counseling (GC) Uptake | 1-month, 6-month follow-up
  GC uptake will be defined as the proportion of participants who undergo genetic counseling within 6 months of the baseline survey (for both the EUC and RA arms). This will be verified through medical record documentation. Self-reported GC will be tracked if verification is not feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Director at Rutgers Cancer Institute
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No